CLINICAL TRIAL: NCT04341363
Title: Follicular Revival in Treatment-resistant Alopecia Areata: Evaluating Use of Micro-needling
Brief Title: Follicular Revival in Androgenic Alopecia: Evaluating Use of Micro-needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000027404
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microneedling (Experimental): Participants with androgenic alopecia will receive microneedling with a tattoo machine.
  Interventions: Device: Tattoo machine

INTERVENTIONS:
Device: Tattoo machine — A SOL Nova Device (brand) tattoo machine will be used to stimulate hair regrowth.

SUMMARY:
The intent of this study is to evaluate the efficacy of microneedling through use of a professional tattoo machine in hair regrowth in patients with androgenic alopecia (AGA) over up to 6 treatments (6 months).

DETAILED DESCRIPTION:
Proposed is an open label trial of tattoo machine microneedling in ten patients with androgenic alopecia. Ten healthy male patients older than 18 years will undergo 6 microneedling sessions. Over the course of six months, subjects will undergo up to six treatment sessions (one session every 30 day). Patients will be evaluated at 8 visits over 8 months with the first visit for screening purposes.

ELIGIBILITY:
Inclusion Criteria:

* Symmetric hair loss from AGA
* Hamilton-Norwood IIIa, III, III vertex, IV, Iva, V with low density hair coverage over majority of alopecic areas
* No or minimal scalp hair regrowth on oral and/or topical minoxidil

Exclusion Criteria:

* Any male with hair loss for other reasons
* Unilateral or asymmetric hair loss
* Hamilton-Norwood I, II, IIa, Va, IV, VII x
* Patients without hair
* Patients with the following who would make poor candidates for microneedling such as skin conditions, diabetes, or history of keloid formation
* Anything additional existing comorbidities that in the opinion of the investigator may cause unnecessary risk for the patient to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, PhD, Principal Investigator — Associate Professor of Dermatology, Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microneedling
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Microneedling
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Total area hair count [Mean (Standard Deviation); unit: hairs per cm^2] | 100.4 (41.4)
SALT Score [Mean (Standard Deviation); unit: percentage of hair loss] | 25.0 (20.2)
Hair Shaft Diameters [Mean (Standard Deviation); unit: micrometer] | 58.0 (15.8)
Number of hair follicles [Mean (Standard Deviation); unit: hair follicles per cm^2] | 96.3 (37.9)
Number of Vellus Hairs [Mean (Standard Deviation); unit: vellus hairs per cm^2] | 13.3 (14.7)
Number of Terminal Hairs [Mean (Standard Deviation); unit: terminal hairs per cm^2] | 87.1 (33.2)

OUTCOME MEASURES:

1. Primary Outcome: Total Area Hair Count
Description: Total number of hairs in an area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: hairs per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 6
hairs per cm^2 | 126.8 (41.7)

2. Secondary Outcome: SALT Score
Description: The Severity of Alopecia Tool measures percentage of scalp hair loss
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of hair loss
Arm/Group | Microneedling
Number analyzed (Participants) | 6
percentage of hair loss | 15.5 (9.7)

3. Secondary Outcome: Hair Shaft Diameter
Description: The diameter of the hair shaft as measured by trichoscopy
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Microneedling
Number analyzed (Participants) | 6
micrometer | 54.4 (8.1)

4. Secondary Outcome: Number of Follicular Units
Description: Number of follicular units with one or more hair follicles over an area of 1cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: follicular units per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 6
follicular units per cm^2 | 108.8 (29.7)

5. Secondary Outcome: Vellus Hairs
Description: Number of vellus hairs over an area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: vellus hairs per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 6
vellus hairs per cm^2 | 18.0 (26.3)

6. Secondary Outcome: Terminal Hairs
Description: Terminal hairs over an area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: terminal hairs per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 6
terminal hairs per cm^2 | 104.3 (21.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Microneedling
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microneedling (N=8)
Subdural hematoma (Vascular disorders) | 1 (1) — Patient slipped on the ice and hit their head (unrelated to study). Patient withdrawn from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04341363/Prot_SAP_000.pdf